CLINICAL TRIAL: NCT02196194
Title: A Prescription-Event Monitoring (PEM) Study of Tiotropium Based on Prescription Data Collected by the Prescription Pricing Authority (PPA) in England for Tiotropium (Spiriva®)
Brief Title: A Prescription-Event Monitoring (PEM) Study of Tiotropium
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.290
Record Dates: First submitted 2014-07-18; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- tiotropium
  Interventions: Drug: Tiotropium

INTERVENTIONS:
Drug: Tiotropium

SUMMARY:
This prescription-event monitoring study was based upon 'event' monitoring and so capable of identifying signals of events that might be associated with the use of tiotropium, which none of the participating general practitioners (GPs) suspected to be an adverse drug reaction. The methodology of this study readily permits follow up of specific events and the obtaining of additional data as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* patients who were prescribed tiotropium

Exclusion Criteria:

* not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with tiotropium
Sampling Method: Non-Probability Sample
Enrollment: 13891 (Actual)
Dates: Start 2002-09; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
incidence density of events | up to sixth month of treatment
  incidence density per 1000 patient-months of treatment